CLINICAL TRIAL: NCT06673693
Title: Neoadjuvant SBRT Sequential Tislelizumab in Locally Advanced Head and Neck Squamous Cell Carcinoma: A Single-Arm Phase II Clinical Study
Brief Title: Tislelizumab Combined With SBRT for the Treatment of Head and Neck Squamous Cell Carcinoma
Acronym: NEOSTART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Chunyan, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-179
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC); HNSCC
Keywords: SBRT; PD-1 antibody; Tislelizumab; Neoadjuvant Therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT combined with PD-1 (Experimental): Week 1: SBRT radiation therapy administered as 24Gy/3f, on days 1, 3, and 5. Weeks 2-5: Tislelizumab 200mg intravenous drip every 3 weeks, for a total of two cycles.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — SBRT
  Other Names: Radiotherapy

SUMMARY:
Exploring the efficacy and safety of Tislelizumab combined with stereotactic body radiation therapy (SBRT) as neoadjuvant treatment for locally advanced head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, initially treated, surgically resectable head and neck squamous cell carcinoma.
* Clinical stage III to IVB (AJCC 8th edition), except HPV-positive oropharyngeal cancer
* Following multidisciplinary discussions involving otolaryngologists and radiation oncologists, the assessment concluded that the tumor is resectable or marginally resectable and suitable for preoperative SBRT
* Karnofsky Performance Status score ≥ 70
* Ages 18 to 70
* The primary organ functions meet the test requirements
* Patients participate voluntarily and sign informed consent forms

Exclusion Criteria:

* Patients previously treated with head and neck surgery were excluded from diagnostic biopsies of primary and regional lymph nodes
* Previous chemotherapy for any reason, or radiotherapy in the head and neck area, or molecular targeted drug therapy; Previously received anti-PD-1, anti-PD-L1, anti-PD-L2 and other drugs or drugs acting on another irritating or co-inhibitory T cell receptor (such as CTLA-4, OX 40, CD137) treatment, or cell biotherapy
* Pregnant or lactating women
* Have had or co-had other malignancies
* The patient also has a serious, uncontrolled illness
* Heart, brain, lung and other important organ function abnormal. Patients with hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg) who cannot be reduced to the normal range by antihypertensive drugs have grade I or above myocardial ischemia or myocardial infarction, arrhythmia, and grade II cardiac insufficiency; Abnormal coagulation function (INR >1.5 or prothrombin time (PT) > ULN+4 seconds or APTT >1.5 ULN), have a tendency to bleed or are receiving thrombolytic or anticoagulant therapy; Have a definite bleeding tendency; Patients with positive urinary protein (urinary protein test 2+ or more, or 24-hour urinary protein quantification >1.0g)
* Glucocorticoid therapy for 30 days prior to initial administration (prednisone equivalent dose > 10mg daily); Have an active autoimmune disease that has required systemic treatment (i.e., disease-modulating drugs, corticosteroids, or immunosuppressive drugs) in the last 2 years
* History of non-infectious pneumonia requiring corticosteroid treatment within 1 year prior to the first dose administration or current presence of interstitial lung disease
* Active infections such as tuberculosis that require systemic treatment
* A known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive)
* Untreated active hepatitis B; Note: Hepatitis B subjects who met the following criteria were also eligible for inclusion: HBV viral load must be <1000 copies /ml (200 IU/ml) prior to initial dosing, and subjects should receive anti-HBV therapy to avoid viral reactivation throughout study chemotherapeutic therapy. Subjects with anti-HBC (+), HBsAg (-), anti-HBS (-) and HBV viral load (-) do not need to receive prophylactic anti-HBV therapy, but need to closely monitor viral reactivation. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection)
* Patients who have a history of psychotropic substance abuse and cannot abstain or have mental disorders
* The investigator determines other circumstances that may affect the conduct of the clinical study and the determination of the study results
* While participating in another therapeutic clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with MPR | From date of first day until the date of obtaining postoperative pathology, assessed up to 4 months
  MPR is defined as < 10% of surviving tumor cells.

SECONDARY OUTCOMES:
Number of Participants with pCR | From date of first day until the date of obtaining postoperative pathology, assessed up to 4 months
  pCR is defined as the absence of viable tumor cells in the postoperative specimen.
Number of Participants with downstaging in Clinical Pathological Staging as assessed by the AJCC 8th Edition Staging System | From date of first day until the date of obtaining postoperative pathology, assessed up to 4 months
  Utilization of the AJCC 8th Edition Staging System for Downstaging from Clinical to Pathological Staging
Median Progression-Free Survival | The time corresponding to a cumulative progression-free survival rate of 50%
  The time corresponding to a cumulative progression-free survival rate of 50%
Median Overall Survival | The time corresponding to a cumulative overall survival rate of 50%
  The time corresponding to a cumulative overall survival rate of 50%. Survival rate is defined as the time from the initiation of the first treatment to death from any cause.
Safety | From the commencement of neoadjuvant therapy until 30 days post-completion
  Assessment of treatment-related adverse events using the Common Terminology Criteria for Adverse Events (CTCAE 5.0) is conducted from the initiation of neoadjuvant therapy through 30 days post-completion of all treatments. Adverse reactions are defined as adverse events related to the investigational drug with a relationship deemed "definitely related/possibly related/unable to determine.
Assessment of Quality of Life | Before treatment, prior to surgery, and within one week after all treatments are completed.
  The Quality of Life (QoL) was assessed at baseline and during follow-up using the European Organization for the Head and Neck Cancer Module (QLQ-H&N35) version 1.0, which represent functions, symptoms, or health conditions. The European Organization for Cancer Research and Treatment QLQ-C30 （EORTC QLQ-C30）: a quality of life instrument for use in international clinical trials in oncology. The evaluation was performed before treatment, 15 minutes after each cycle of chemotherapy, and 3 and 6 months after the end of treatment. A total of 30 items are included. Each item is graded from 1 to 4, except for items 29 and 30, indicating not at all, a little, quite a bit, and very much, with higher scores indicating poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No